CLINICAL TRIAL: NCT02899273
Title: Perception of Children With Visible Untreated and Treated Caries
Acronym: ECC-ET
Status: Completed | Type: Observational
Sponsor: University of Göttingen (Other)
Collaborators: Stiftung Universität Hildesheim (Unknown)
Responsible Party: Principal Investigator, Claudia Tschammler, Postdoctoral Research Fellow, University of Göttingen
Other Study IDs: 36/2/16
Record Dates: First submitted 2016-08-26; First posted 2016-09-14 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Dental Caries
Keywords: Early Childhood Caries; eye-tracking; children; dentistry; face perception
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dentistry students: Dentistry students of the University of Göttingen
- Psychology students: Psychology students of the University of Hildesheim

SUMMARY:
In Germany about 5 to 20% of children suffer from early childhood caries (ECC). Preceding results of eye-tracking-studies on the perception of patients with unilateral cleft and patients with severe orthognathic malocclusion let us assume that caries and missing teeth might influence the observer's focus. The aim of this study is to test the hypothesis that the faces of patients with ECC and patients with signs of dental treatment (crown, gap etc.) are contemplated differently from and assessed more negatively than healthy patients. Particular attention should be paid to potential differences between the findings of the two observer-groups (medical laypersons/ dental students).

DETAILED DESCRIPTION:
In Germany about 5 to 20% of children suffer from early childhood caries (ECC). Resulting in complications like damages of the permanent teeth, pain and developmental disorder of the affected jaw, ECC might additionally lead to social exclusion. Previous eye-tracking-studies about the perception of patients with unilateral cleft and patients with severe orthognathic malocclusion demonstrated that these variations are transferring the observer's focus from the eyes and nose to the affected region. The aim of this study is to test the hypothesis that the faces of patients with ECC and patients with signs of dental treatment (crown, gap etc.) are contemplated differently from and assessed more negatively than healthy patients. Particular attention should be paid to potential differences between the findings of the two observer-groups (medical laypersons/ dental students).

ELIGIBILITY:
Inclusion Criteria:

* healthy
* student of the University of Göttingen or Hildesheim
* age ≥ 18 years
* people who agreed to participate in the study
* right-hander

Exclusion Criteria:

* missing agreement to participate in the study
* missing cooperation,
* age < 18 years
* left-hander
* wearer of glasses
* people with severe systemic diseases, especially states with associated temporary or permanent restriction of immune status
* people with severe mental illness who have altered perception or neurophysiological stimulus processing.
* people who take regularly or at the time of the study drug or drugs that altered a perception or neurophysiological stimulus processing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-12-08 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
The first fixation on one of both pictures will be measured | 3 sec
  both pictures: a) emotional, b) neutral

SECONDARY OUTCOMES:
First fixation of one of three areas of interest will be measured | 300 msec
  areas of interest: a) eyes, b) nose, c) mouth
Fixation time and fixation number of areas of interest will be measured | 2 sec
  areas of interest: a) eyes, b) nose, c) mouth
Are the pictures different in valence, arousal, attractiveness | 30 min
  Questionnaire:
  1. How pleasant this stimulus is for you? (9 point scale: 1 negative - 9 positive)
  2. How exciting is this stimulus to you? (9 point scale: 1 low - 9 high) 3 How attractive is this appeal to you? (9 point scale: 1 unattractive - 9 attractive) Self-Assessment-Manikin scales

CONTACTS AND LOCATIONS:
Overall Officials: Annette Wiegand, Prof. Dr., Study Director — Dept. of Prev. Dentistry, Periodontology and Cariology, University Medical Center Göttingen, Germany; Kristian Folta-Schoofs, Prof. Dr., Study Chair — Dep. of Psychology, Stiftung Universität Hildesheim, Germany
Locations (2):
- Germany (2):
  - Department of Preventive Dentistry, Periodontology and Cariology, University Medical Center Goettingen, Germany, Göttingen, Lower Saxony
  - Cognitive Neuroscience Lab, Institute of Psychology, University of Hildesheim Hildesheim, Germany, Hildesheim, Lower Saxony

IPD SHARING:
Plan to Share IPD: Undecided